CLINICAL TRIAL: NCT02626585
Title: The Effect of Postrhinoplasty Taping on Postoperative Edema and Nasal Draping
Acronym: PRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Berke Özücer, Otorhinolaryngologist, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BezmialemVU-BO-PRT
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Nasal Deformity; Edema; Rhinoplasty
Keywords: rhinoplasty; postrhinoplasty taping; edema; draping; postoperative edema; nasal skin thickness; supratip fullness; postoperative swelling
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Control group (n=20): Following removal of nasal cast on postoperative first week, no additional taping was applied to this group.
- 2-weeks of PRT (Experimental): 2-weeks of PRT (n=17): Following removal of nasal cast on postoperative first week, 2 weeks of additional postrhinoplasty taping was applied to this group (form 1st to 3rd week).
  Interventions: Procedure: Postrhinoplasty taping
- 4-weeks of PRT (Experimental): 4-weeks of PRT (n=20): Following removal of nasal cast on postoperative first week, 4 weeks of additional postrhinoplasty taping was applied to this group (form 1st to 5th week).
  Interventions: Procedure: Postrhinoplasty taping

INTERVENTIONS:
Procedure: Postrhinoplasty taping — Postrhinoplasty taping is commonly applied by rhinoplasty surgeons. Following rhinoplasty the nose is generally taped and a (thermoplastic) nasal cast is applied on top of this to make sure the final form of the nose is protected. Postoperatively, this cast is removed at some point. After this, some of the surgeons prefer to tape the nose with nasal tapes such as Micropore (3M) etc. Postrhinoplasty taping is the term used for this. The nose is (generally) taped horizontally with 1/2 inch wide tapes. This is done superiorly from radix to inferiorly to nasal tip. The idea is to compress the nose and to cover it. The duration of postrhinoplasty taping differs according to the preference of the surgeon and the patient
  Arms: 2-weeks of PRT; 4-weeks of PRT

SUMMARY:
The purpose of this study was to investigate the effectiveness of postrhinoplasty taping. The effectiveness was evaluated with Ultrasonography and skin envelope thickness was prospectively measured for analysis.

DETAILED DESCRIPTION:
All patients were informed individually about the procedures and written informed consent was obtained before the study. Undergoing primary open approach reduction rhinoplasty and receiving osteotomies with lateral guarded osteotomes was an inclusion criteria for the study. Fifty-seven consecutive primary open approach rhinoplasty patients that referred to our tertiary reference center were enrolled in the study. Patients were appointed to either the control, 2-week PRT or 4-week PRT group in a randomized-consecutive fashion. External thermoplastic splint was removed at the end of first postoperative week. Patients in the control group were not subjected to further nasal taping after cast removal. All patients in 2-week (from first to third week) and 4-week (from first to fifth week) PRT groups received taping during their allocated time in addition to one week with external nasal splint. These two groups were provided with 1/2-inch wide tan-colored hypoallergenic 3M™ Micropore™ Surgical Tapes (3M, St Paul, Minnesota). Each volunteer was individually shown how and given instructions regarding PRT.

Nasal swelling of the patients were evaluated individually with a 7.5 mHz linear ultrasound (US) probe: small amount of ultrasonic gel was used to scan the skin in a noncontact mode to prevent distortion of nasal anatomy from transducer pressure. The examiner did not have access to the results of the previously obtained measurements in order to prevent measurements from being contaminated. Measurements were carried out on four different points: nasion, rhinion, supratip and tip and from these four measurements, mean nasal skin thickness (MNST) was calculated.

Subjects in each group were sorted, based on the baseline MNST measurement, consecutively from lowest to highest; half of the patients with higher MNST measurements were categorized as 'thick skinned' and the other half was categorized as 'thin skinned'. The electronic caliper of the machine measured the perpendicular distance from the outer epidermal surface to the underlying cartilage on the 2-dimensional B-mode image (Capasee II Ultrasound, Toshiba Medical Systems, Tustin, California). US measurements were carried out five times for each individual subject: preoperatively; at the end of first, third and fifth postoperative weeks; and sixth postoperative month. Measurements were carried out mainly in the morning to avoid the effect of diurnal variation on the dermal edema.

Surgical Technique All of the patients were operated with open approach rhinoplasty under general anesthesia. All patients underwent rhinoplasty due to cosmetic and functional purposes. All cases were distributed evenly between the surgeons (BO, YSY, BV, ST). Supraperichondrial and subperiosteal dissection plane was the preferred plane of dissection in all the cases. Surgical operation was mainly reduction rhinoplasty and comprised of dorsal reduction and bilateral lateral osteotomies. All lateral osteotomies were carried out intranasally with guarded curved lateral osteotomes. Incision-to-closure operative duration was recorded for each patient. All subjects were routinely administered 0.1mg/kg dexamethasone during the operation. All cases were applied with internal splints, taped with 3M micropores and casted with external thermoplastic splints at the end of the operation. Postoperative suggestions, orders and medications were identical for all groups. Patients were discharged from the hospital on first postoperative day. All subjects were called back on the end of first postoperative week for removal of external nasal packing.

Statistical Analysis Statistical data were analysed using SPSS 20.0 (SPSS, Chicago,IL). All values were calculated and stated in descriptive statistics as mean±Standard deviation unless otherwise stated. ANOVA was used for comparison of means. Repeated ANOVA was used for each patient where the repeated factor was the ultrasonographic measurements (preoperative, first postoperative week, third postoperative week, fifth postoperative week and sixth postoperative month). Significant results of repeated ANOVA test were further analysed via pairwise comparison with Bonferroni correction. Correlation analysis was carried out with Pearson correlation analysis. Values of p<0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* primary open approach rhinoplasty under general anesthesia
* bilateral lateral osteotomies

Exclusion Criteria:

* revision cases
* abnormal haemostatic parameters
* drug history of decongestant or cortisone

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in nasal skin thickness (for rhinion, radix, supratip and tip) | preoperative, postoperative 1st, 3rd and 5th week, postoperative 6th month
  measured with Ultrasonography

SECONDARY OUTCOMES:
Duration of Operation | Intraoperative
  (minutes)(incision to closure duration)

CONTACTS AND LOCATIONS:
Overall Officials: Berke Ozucer, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hafezi F, Naghibzadeh B, Nouhi A. Management of the thick-skinned nose: A more effective approach. Ann Otol Rhinol Laryngol. 2006 Jun;115(6):444-9. doi: 10.1177/000348940611500608. PMID 16805376
- [Background] Guyuron B, DeLuca L, Lash R. Supratip deformity: a closer look. Plast Reconstr Surg. 2000 Mar;105(3):1140-51; discussion 1152-3. doi: 10.1097/00006534-200003000-00049. PMID 10724276
- [Background] Rees TD. An aid to the treatment of supratip swelling after rhinoplasty. Laryngoscope. 1971 Feb;81(2):308-11. doi: 10.1288/00005537-197102000-00011. No abstract available. PMID 5544202
- [Background] Hoefflin SM. Postoperative nighttime nasal taping to decrease swelling. Plast Reconstr Surg. 1989 Aug;84(2):375. doi: 10.1097/00006534-198908000-00057. No abstract available. PMID 2748764
- [Background] Vega-Villasante P, Covarrubias H. A new splint for the nasal tip. Plast Reconstr Surg. 1995 Jul;96(1):189-93. doi: 10.1097/00006534-199507000-00029. PMID 7604101
- [Background] Belek KA, Gruber RP. The beneficial effects of postrhinoplasty taping: fact or fiction? Aesthet Surg J. 2014 Jan 1;34(1):56-60. doi: 10.1177/1090820X13515879. PMID 24396072
- [Derived] Ozucer B, Yildirim YS, Veyseller B, Tugrul S, Eren SB, Aksoy F, Uysal O, Ozturan O. Effect of Postrhinoplasty Taping on Postoperative Edema and Nasal Draping: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2016 May 1;18(3):157-63. doi: 10.1001/jamafacial.2015.1944. PMID 26914594